CLINICAL TRIAL: NCT01383083
Title: Effects of Iloprost Treatment in Adult Patients With Pulmonary Arterial Hypertension Related to Congenital Heart Disease (Eisenmenger Physiology): Safety, Tolerability, Clinical, and Hemodynamic Effect.
Brief Title: Effects of Iloprost Treatment in Adult Patients With Pulmonary Arterial Hypertension Related to Congenital Heart Disease
Acronym: EIGER
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Maryknoll Medical Center (Other)
Collaborators: Pusan National University Hospital (Other); Inje University (Other); Yeungnam University Hospital (Other)
Responsible Party: Kyoung Im Cho, Maryknoll Medical Center
Other Study IDs: EIGER2011
Record Dates: First submitted 2010-11-29; First posted 2011-06-28 (Estimated); Last update posted 2011-06-28 (Estimated); Status verified 2010-11

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: Pulmonary arterial hypertension; Congenital heart disease; Eisenmenger physiology
MeSH Terms: conditions — Pulmonary Arterial Hypertension; Heart Defects, Congenital

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- iloprost: In the adult patient group, iloprost acceptable target dose is 2.5 ug 4-6 times/day according to the patient's compliance. Because of the concern of safety and tolerability, during the first 4 weeks of treatment, patients receive 2.5 ug twice daily. After 4 weeks, this is increased to the target dose, if iloprost is well tolerated.

SUMMARY:
The prevalence of PAH associated with congenital systemic-to-pulmonary shunts in Western countries has been estimated to range between 1.6 and 12.5 cases per million adults, with 25-50% of this population affected by Eisenmenger's syndrome. The rarity of this syndrome, combined with its complex pathophysiology, account for the insufficient understanding of the principles underlying its proper treatment.Recent decades have seen developments in pulmonary hypertension pathophysiology which have led to the introduction of new groups of drugs: prostacycline analogs (Epoprostenol, Treprostinil, Beraprost, Illoprost), phosphodiesterase inhibitors (Sildenafil, Tadalafil), endothelin receptor antagonists (Bosentan, Sitaxantan, Ambrisentan) and nitric oxide. These drugs should be administered to patients in III-IV NYHA class. Despite successful early results, the therapeutic effect on patients with Eisenmenger syndrome has not been conclusively established The treatment strategy for patients with PAH associated with congenital systemic-to-pulmonary shunts and, in particular, those with Eisenmenger's syndrome is based mainly on clinical experience rather than being evidence based. Although Eisenmenger's syndrome is uncurable disease, the survival rate is relatively higher than primary PAH, and the patients with Eisenmenger's syndrome are relatively younger group. So the improvement of exercise tolerance and quality of life is very important. Several randomized controlled trial reported favourable short- and long-term outcomes of treatment with the orally active dual endothelin receptor antagonist bosentan in patients with Eisenmenger's syndrome. However, there was scare data of outcomes of treatment with the inhaled iloprost in patients with Eisenmenger's syndrome. In Korea, most of patients with Eisenmenger's syndrome are treated with conservative therapy instead of administration of PAH-specific drug, because of lack of clinical experience. Moreover, oral agent such as bosentan, sidenafil is preferred than iloprost becase of more evidence and convenience. Our therapeutic efforts should be directed mainly towards preventing complications. As a rule, we should avoid agents with no established therapeutic efficacy and try to alleviate symptoms without any additional risk, so as not to disrupt the existing clinical balance.

In this study, we investigate to know the clinical benefit of iloprost on patients with Eisenmenger's syndrome by the use of functional and hemodynamic parameters, which would add the evidence of PAH-specific agents on the Eisenmenger's syndrome

DETAILED DESCRIPTION:
A large proportion of patients with congenital heart disease (CHD), in particular those with relevant systemic-to-pulmonary shunts, will develop pulmonary arterial hypertension (PAH) if left untreated. Persistent exposure of the pulmonary vasculature to increased blood flow, as well as increased pressure, may result in pulmonary obstructive arteriopathy, which leads to increased pulmonary vascular resistance that, if it approaches or exceeds systemic resistance, will result in shunt reversal. Eisenmenger's syndrome, the most advanced form of PAH associated with CHD, is defined as CHD with an initial large systemic-to-pulmonary shunt that induces severe pulmonary vascular disease and PAH, with resultant reversal of the shunt and central cyanosis. The histopathological and pathobiological changes seen in patients with PAH associated with congenital systemic-to-pulmonary shunts, such as endothelial dysfunction of the pulmonary vasculature, are considered similar to those observed in idiopathic or other associated forms of PAH.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with Eisenmenger syndrome are clinically stable and in World Health Organization functional class (WHO class) III or worse are selected for treatment.
2. Eisenmenger syndrome is diagnosed echocardiographically as right-to-left shunting through the shunt defect.
3. To exclude other causes of PAH, lung function tests (spirometry, forced expiratory volume in 1 second, and forced vital capacity)are obtained.

Exclusion Criteria:

1. Patients with severe left ventricular dysfunction and/or pulmonary venous congestion (measured invasively or assessed echocardiographically) are excluded.
2. Patients with obstruction of the right ventricular outflow tract, pulmonary valve, or pulmonary arteries or patients on prostacyclin, glibenclamide, or cyclosporine treatment were excluded.
3. Patients with contraindication to Ventavis;

   * Hypersensitive to Ventavis
   * High risk of bleeding, which can be increased by use of Ventavis (e.g. active peptic ulcer, trauma, intracranial hemorrhage)
   * Severe coronary disease, unstable angina, history of Acute myocardial infarction within 6 months, uncompensated heart failure not under close medical monitoring, severe arrhythmia, suspected pulmonary congestion, cerebrovascular disease within 3 months (e.g. transient ischemic attack, stoke)
   * pulmonary hypertension due to venous occlusive disease
   * valvular defect with dysfunction of cardiac muscle, which is independent of pulmonary hypertension
   * pregnancy, women with high probability of pregnancy, breast feeding
   * renal failure (creatinine clearance <30mL/min)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PAH associated with congenital systemic-to-pulmonary shuntand treated with iloprost for pulmonary hypertension
  : patients with PAH associated with corrected and uncorrected congenital systemic-to-pulmonary shunts and Eisenmenger's syndrome are included
Sampling Method: Probability Sample
Enrollment: 42 (Estimated)
Dates: Start 2010-11; Primary Completion 2011-06 (Estimated); Study Completion 2012-11 (Estimated)

PRIMARY OUTCOMES:
Pulmonary Vascular Resistance | Change from Baseline in PVR at 24 weeks
  To identify hemodynamic benefit and safety of 24 weeks treatment with iloprost on patients with Eisenmenger's syndrom

SECONDARY OUTCOMES:
Assessment of quality of life | Change from Baseline in QoL at 24 weeks
  To investigate the change of quality of life(SF-12) after 24 weeks treatment with iloprost
Exercise capacity | Change from baseline in exercise capacity at 24 weeks
  To investigate the change of exercise capacity(6-minute walking test) after 24 weeks treatment with iloprost

CONTACTS AND LOCATIONS:
Overall Officials: Kyoung Im Cho, MD, Principal Investigator — Maryknoll General Hospital